CLINICAL TRIAL: NCT02569606
Title: Transfusion and Coagulation Management in Trauma Patients After the Introduction of a Coagulation Algorithm
Status: Completed | Type: Observational
Sponsor: Donat R. Spahn (Other)
Collaborators: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor-Investigator, Donat R. Spahn, Head of Institut of Anesthesiology University Hospital Zurich, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: ZH 2015 - 0309
Record Dates: First submitted 2015-09-30; First posted 2015-10-07 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Hemorrhage
Keywords: consumption of blood; consumption of coagulation products; coagulation algorithm; trauma related transfusion
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Timeframe 2005 - 2007: Data of timeframe 2005 up to 2007 will be included
- Timeframe 2012 - 2014: Data of timeframe 2012 up to 2014 will be included

SUMMARY:
Comparison of the consumption of blood and coagulation products (packed red blood cells, fresh frozen plasma, platelet concentrates, fibrinogen, coagulation factor concentrates, coagulation factor XIII, activated factor VII, van Willebrand factor and antifibrinolytics) before and after the introduction of a designated trauma related transfusion and coagulation algorithm.The periods 2005-2007 (before) and 2012-2014 (after) the introduction are reviewed. Two level-1 trauma centers in Switzerland (Hospital Lucerne, University Hospital Zurich) are included in the study. Predicted probability of a massive transfusion by the trauma associated acute hemorrhage score (TASH)is correlated with the actual rate.

DETAILED DESCRIPTION:
Trauma is one of the leading causes of death worldwide. After death due to direct craniofacial injury, exsanguination is the next major cause for trauma mortality.

After initial pre-hospital treatment the patient is admitted to the hospital. If multiple injuries are present the patient is transferred to a specialized trauma center.

Besides surgical treatment, the patient needs stabilization of the vital functions by the Anesthesiologist. Due to loss of blood volume, dilution of the circulatory blood volume and pathological activation of coagulation/fibrinolysis, trauma induced coagulopathy (TIC) is initiated. This needs to be treated and avoided whenever possible.

Transfusion of allogeneic blood and coagulation product itself leads to an increased morbidity and mortality. Infectious and immunologic reactions account for that phenomenon.

This led to a paradigm change in the therapy of TIC. In 2009 a new coagulation factor based coagulation algorithm was introduced in the Hospital Lucerne and the University Hospital in Zurich / Switzerland. With the help of point of care coagulation measurement, tailored coagulation factor based coagulation management and avoidance of allogeneic blood products was initiated.

The investigators now want to analyze the impact of the coagulation algorithm by comparing the periods before and after the introduction of the algorithm.

The consumption of blood and coagulation products (packed red blood cells, fresh frozen plasma, platelet concentrates, fibrinogen, coagulation factor concentrates, coagulation factor XIII, activated factor VII, van Willebrand factor and antifibrinolytics) before and after the introduction of a designated trauma related transfusion and coagulation algorithm will be recorded and compared. The periods 2005-2007 (before) and 2012-2014 (after) the introduction are reviewed. Predicted probability of a massive transfusion by the TASH score (trauma associated acute hemorrhage) is correlated with the actual rate.

ELIGIBILITY:
Inclusion Criteria:

* male and female trauma patients
* admitted to the University hospital of Zurich or the Hospital of Lucerne, Switzerland
* injury severity score >= 16
* time period 2005-2007 and 2012-2014

Exclusion Criteria:

* incomplete data
* denial of informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients with an injury severity score (ISS) >15 treated in University Hospital Zurich or Lucerne hospital during 2005 to 2007 and 2012 to 2014
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Comparison the consumption of red blood cells, fresh frozen plasma and platelets in the treatment period by the Anaesthesist and after 24/48 hours before (2005-2007) and after (2012-2014) launching the coagulation algorithm. | up to 48 hours
  The coagulation algorithm was launched in 2010. To show the difference in transfusion and administration of coagulation products prior and after the changes of coagulation algorithm the probability of massive transfusion (TASH Score) will be compared with the actual rate. The TASH Score is the most precise predictive probability of a massive transfusion. Data of approximately 1800 participants will be compared.
Comparison of the rate of massive transfusion in reality with the predicted rate (by TASH) score. | up to 48 hours
  Massive transfusion (>10 units of blood) can be predicted on the base of patient and trauma epidemiology. The investigator compares the actual rate in the institution with the rate predicted by the score.

SECONDARY OUTCOMES:
Comparison of the predicted mortality (TRISS/RISC2) with the actual rate | up to 30 days
  TRISS is a common Score and is a comparative value for trauma mortality outcome. The investigators want to show the benefit of launched coagulation algorithm in mortality after severe trauma.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Lucerne Kantonssital, Lucerne
  - University Hospital Zurich, Zurich